CLINICAL TRIAL: NCT04171765
Title: A Phase II, Randomized, Parallel-Group, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of BFKB8488A Compared With Placebo in Patients With Non-Alcoholic Steatohepatitis
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of BFKB8488A Compared With Placebo in Participants With Non-Alcoholic Steatohepatitis
Acronym: BANFF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to strategic business reasons.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GC41033
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants will receive a fixed dose of placebo matched to BFKB8488A.
  Interventions: Drug: Placebo
- Fixed Dose: BFKB8488A Dose A (Experimental): Participants will receive BFKB8488A.
  Interventions: Drug: BFKB8488A
- Fixed Dose: BFKB8488A Dose B (Experimental): Participants will receive BFKB8488A.
  Interventions: Drug: BFKB8488A
- Fixed Dose: BFKB8488A Dose C (Experimental): Participants will receive BFKB8488A.
  Interventions: Drug: BFKB8488A

INTERVENTIONS:
Drug: Placebo — Participants will receive subcutaneous (SC) placebo matched to BFKB8488A.
  Arms: Placebo
Drug: BFKB8488A — Participants will receive subcutaneous (SC) BFKB8488A.
  Arms: Fixed Dose: BFKB8488A Dose A; Fixed Dose: BFKB8488A Dose B; Fixed Dose: BFKB8488A Dose C

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacokinetics of BFKB8488A compared to placebo in participants with non-alcoholic steatohepatitis (NASH).

ELIGIBILITY:
Inclusion Criteria

* Confirmed diagnosis of NASH as documented through liver biopsy performed no more than 6 months before randomization, defined according to NASH CRN criteria along with a NASH CRN fibrosis score between F2 and F3
* Hepatic steatosis on MRI (>= 8% average PDFF) prior to randomization

Exclusion Criteria

* History of any liver disease other than NASH, except for resolved, self-limited illnesses such as Hepatitis A or E, and previous Hepatitis C
* Weight gain > 10% or loss > 5% within 3 months prior to randomization
* History of liver transplantation
* Current or history of significant alcohol consumption

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (53):
- United States (39):
  - Cullman Clinical Trials, Cullman, Alabama
  - Arizona Liver Health - Chandler, Chandler, Arizona
  - Arizona Liver Health - Tucson, Tucson, Arizona
  - Orange Grove Family Practice, Tucson, Arizona
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Gregory Wiener, MD, Chula Vista, California
  - Community Cancer Institute (CCI), Fresno, California
  - National Research Inst., Los Angeles, California
  - Conquest Clinical Research, Orange, California
  - UC San Diego Airway Research and Clinical Trials Center, San Diego, California
  - National Research Institute - Panorama City, Santa Monica, California
  - South Denver Gastroenterology, Englewood, Colorado
  - Excel Medical Research, Boca Raton, Florida
  - Premier Research Associate, Inc, Miami, Florida
  - Covenant Research, Sarasota, Florida
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Grand Teton Research Group, PLLC, Idaho Falls, Idaho
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Avant Research Associates, LLC, Crowley, Louisiana
  - Walter Reed Army Medical Center, Bethesda, Maryland
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - Kansas City Research Institute, LLC, Kansas City, Missouri
  - Amici Clinical Research, Raritan, New Jersey
  - Duke Medical Center; Gen Clinic Research Ctr, Durham, North Carolina
  - Wexner Medical Center; Ohio State University; Investigational Drug Services; Pharmacy Department, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Pinnacle Clinical Research - Austin, Austin, Texas
  - Texas Digetive Disease Consultants - Austin, Cedar Park, Texas
  - Liver Institute at Renaissance, Edinburg, Texas
  - South Texas Research Institute, Edinburg, Texas
  - Texas Digestive Disease Consultant - Ft Worth (TDDC - Ft Worth), Fort Worth, Texas
  - Liver Associates of Texas - Houston, Houston, Texas
  - Quality Research Inc, San Antonio, Texas
  - American Research Corporation Inc., San Antonio, Texas
  - Clinical Trials of Texas, Inc, San Antonio, Texas
  - Pinnacle Clinical Research - San Antonio, San Antonio, Texas
  - Texas Digestive Disease Consultants - San Marcos, San Marcos, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Hunter Holmes McGuire V.A. Medical Center, Richmond, Virginia
- Belgium (3):
  - Hospital Erasme, Brussels
  - Antwerp University Hospital, Edegem
  - Universitair Ziekenhuis Gent, Ghent
- France (5):
  - CHU Hopitaux de Bordeaux, CHU Hopitaux de Bordeaux
  - Hospices Civils de Lyon, Lyon
  - CHU de Nice, Nice
  - Hopital Pitie-Salpetriere APHP, Paris
  - Hôpital d'Enfants, Service d?onco-hématologie pédiatrique, Vandœuvre-lès-Nancy
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universtiario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia; Servicio de Anatomia Patologica, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe; Servicio de Neurología, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo by subcutaneous (SC) injection every two weeks (Q2W) for 52 weeks.
- Fixed Dose 50 mg: Participants received 50 mg of SC fazpilodemab (BFKB8488A) Q2W for 52 weeks.
- Fixed Dose 75 mg: Participants received 75 mg of SC fazpilodemab (BFKB8488A) Q2W for 52 weeks.
- Fixed Dose 100 mg: Participants received 100 mg of SC fazpilodemab (BFKB8488A) Q2W for 52 weeks.
Period: Overall Study
Arm/Group | Placebo | Fixed Dose 50 mg | Fixed Dose 75 mg | Fixed Dose 100 mg
Started | 13 | 11 | 11 | 11
Completed | 8 | 9 | 7 | 6
Not Completed | 5 | 2 | 4 | 5
Not completed — Adverse Event | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 2 | 2
Not completed — Week 58 visit missed | 0 | 0 | 1 | 0
Not completed — Study terminated by sponsor | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fixed Dose 50 mg | Fixed Dose 75 mg | Fixed Dose 100 mg | Total
Number analyzed (Participants) | 13 | 11 | 11 | 11 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.4 (9.6) | 57.4 (10.0) | 55.4 (8.2) | 51.9 (14.8) | 53.0 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 6 | 24
  Male | 7 | 5 | 5 | 5 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 3 | 5 | 20
  Not Hispanic or Latino | 6 | 6 | 8 | 6 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 2
  White | 13 | 10 | 9 | 10 | 42
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With NASH Resolution on Overall Histopathological Reading Without Worsening of Fibrosis at Week 52
Description: Resolution of non-alcoholic steatohepatitis (NASH) is defined as a non-alcoholic fatty liver disease activity score (NAS) of 0-1 for inflammation, 0 for ballooning, and any value for steatosis as determined by a central reader. Worsening of fibrosis is defined as any increase in NASH Clinical Research Network (CRN) fibrosis stage as determined by a central reader.
Time Frame: Week 52
Population: The modified intent-to-treat (mITT) population was defined as all randomly allocated participants who received at least one dose of study drug or placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo | Fixed Dose 50 mg | Fixed Dose 75 mg | Fixed Dose 100 mg
Number analyzed (Participants) | 6 | 8 | 7 | 6
Percentage of Participants | 16.7 [0.00 to 54.82] | 37.5 [0.00 to 77.30] | 14.3 [0.00 to 47.35] | 33.3 [0.00 to 79.39]

2. Secondary Outcome: Change From Baseline in Hepatic Fat Fraction as Assessed by Magnetic Resonance Imaging-Derived Proton Density Fat Fraction (MRI-PDFF) at Week 52
Time Frame: Baseline, Week 16, Week 52
Population: The mITT population was defined as all randomly allocated participants who received at least one dose of study drug or placebo.
Measure: Mean (Standard Deviation); unit: percentage of hepatic fat fraction
Arm/Group | Placebo | Fixed Dose 50 mg | Fixed Dose 75 mg | Fixed Dose 100 mg
Number analyzed (Participants) | 13 | 11 | 11 | 11
percentage of hepatic fat fraction
  Baseline | 20.15 (6.35) | 20.67 (6.05) | 19.30 (3.99) | 18.12 (7.70)
  Week 16 change from baseline: number analyzed (Participants) | 10 | 8 | 9 | 8
  Week 16 change from baseline | -3.47 (2.28) | -8.20 (8.58) | -2.23 (9.05) | -10.25 (4.76)
  Week 52 change from baseline: number analyzed (Participants) | 7 | 7 | 7 | 6
  Week 52 change from baseline | -4.46 (6.23) | -2.50 (8.13) | -3.46 (11.57) | -3.53 (6.54)

3. Secondary Outcome: Proportion of Participants With Improvement in Liver Histology From Baseline and no Worsening of Fibrosis at Week 52
Time Frame: Week 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Fixed Dose 50 mg | Fixed Dose 75 mg | Fixed Dose 100 mg
Number analyzed (Participants) | 6 | 8 | 7 | 6
Percentage of participants | 16.7 [0.00 to 54.82] | 37.5 [0.00 to 77.30] | 42.9 [0.00 to 86.66] | 33.3 [0.00 to 79.39]

4. Secondary Outcome: Proportion of Participants With Improvement in Liver Fibrosis of at Least One Stage, as Defined by NASH Clinical Research Network (CRN), and no Worsening of NASH at Week 52
Time Frame: Week 52
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Fixed Dose 50 mg | Fixed Dose 75 mg | Fixed Dose 100 mg
Number analyzed (Participants) | 6 | 8 | 7 | 6
Percentage of participants | 16.7 [0.00 to 54.82] | 25.0 [0.00 to 61.26] | 28.6 [0.00 to 69.18] | 16.7 [0.00 to 54.82]

ADVERSE EVENTS:
Time Frame: Through Week 58
Groups:
- Fixed Dose-50mg BFKB8488A: Participants received 50 mg of SC fazpilodemab (BFKB8488A) Q2W for 52 weeks.
- Fixed Dose-75mg BFKB8488A: Participants received 75 mg of SC fazpilodemab (BFKB8488A) Q2W for 52 weeks.
- Fixed Dose-100mg BFKB8488A: Participants received 100 mg of SC fazpilodemab (BFKB8488A) Q2W for 52 weeks.
Arm/Group | Placebo | Fixed Dose-50mg BFKB8488A | Fixed Dose-75mg BFKB8488A | Fixed Dose-100mg BFKB8488A
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/11 | 1/11 | 0/11
Other Adverse Events (participants affected / at risk) | 9/13 | 11/11 | 9/11 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Fixed Dose-50mg BFKB8488A (N=11) | Fixed Dose-75mg BFKB8488A (N=11) | Fixed Dose-100mg BFKB8488A (N=11)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Fixed Dose-50mg BFKB8488A (N=11) | Fixed Dose-75mg BFKB8488A (N=11) | Fixed Dose-100mg BFKB8488A (N=11)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (5) | 3 (4) | 4 (4)
Duodenal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (5) | 1 (1) | 5 (12)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (3) | 2 (2)
Administration site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Administration site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Early satiety (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 5 (5) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cortisol free urine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insulin-like growth factor decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Emotional disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast calcifications (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal valve collapse (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Because the study was terminated early, the interpretation of its data is limited, and early dropout may confound the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT04171765/Prot_SAP_000.pdf